CLINICAL TRIAL: NCT06012253
Title: The Effect of Home-Based Walking Program on Peripheral Neuropathy, Fatigue and Quality of Life in Patients Receiving Taxane and Platinum-Based Chemotherapy
Brief Title: The Effect of Home-Based Walking Program on Peripheral Neuropathy, Fatigue and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University Hospital (Other)
Responsible Party: Principal Investigator, Hava Kara, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: "70904504/376"
Record Dates: First submitted 2023-08-19; First posted 2023-08-25 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chemotherapeutic Toxicity
Keywords: Home-based walking program; Chemotherapy; Cancer; Peripheral neuropathy; Fatigue; Quality of life; Nurse
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases; Fatigue

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial consisting of two groups: experimental and control
Who Masked: Participant, Outcomes Assessor
Masking Description: Single Blind (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Based Walking Program (Experimental): Effect of home-based walking program on peripheral neuropathy, fatigue and quality of life
  Interventions: Other: Home Based Walking Program
- Control group (No Intervention): The control group will be given the "Ministry of Health Physical Activity Guidelines".Routine care.

INTERVENTIONS:
Other: Home Based Walking Program — The intervention group will be applied to "Home Based Walking Program". It was aimed that the patients should do at least 150 minutes of moderate-intensity physical exercise per week for up to 8 weeks. The content of the program includes a walking information booklet (information notes, activity chart and obstacle avoidance form), exercise diary, face-to-face-telephone counseling, sending text messages, prepared in line with international guides. It was planned to give weekly counseling to the patients included in the intervention group for an 8-week period.
  Arms: Home Based Walking Program

SUMMARY:
The study aims to evaluate the effect of home-based walking program on peripheral neuropathy, fatigue and quality of life in patients receiving taxane and platinum-based chemotherapy.

DETAILED DESCRIPTION:
The study was designed as a randomized controlled trial. This study will be carried out with a total of 88 cancer patients receiving taxane and platinum-based chemotherapy, 44 of whom were in the intervention group and 44 in the control group, whose treatment was started in Akdeniz University Hospital."Home Based Walking Program" will be applied to the patients in the intervention group for 8 weeks.Within the scope of the Home-Based Walking Program, face-to-face patient education, patient education booklet, sending text messages, face-to-face and telephone counseling were planned.

Patient Identification Form, International Physical Activity Questionnaire (IPAQ- Short Form), National Cancer Institute (NCI) -CTCAE v5.0 Toxicity Criteria, Cancer Fatigue Scale, EORTC QLQ-CIPN20 (Quality of Life Chemotherapy-Induced Peripheral Neuropathy) and EORTC QLQ-C30 (Quality of Life Scale), Interview Form will be used to collect data.

ELIGIBILITY:
İnclusion Criteria

* 18 Years and older (Adult, Older Adult )
* Turkish speaking-understanding ability and literate.
* Orientation (person, place, time)
* Receiving taxane and platinum-based chemotherapy treatment (monotherapy or combined).
* Receiving chemotherapy treatment for the first time.
* The primary medical diagnosis is cancer (breast cancer, colorectal cancers and other cancers).
* Not having health problems that prevent walking.
* Agreeing to participate in the research.

Exclusion Criteria

* Being bone and brain metastases
* Being peripheral neuropathy due to reasons other than chemotherapy (such as chronic disease, diabetes mellitus, nutritional disorders)
* Skin sensitivity on the hands and feet
* Having cardiovascular, pulmonary, musculoskeletal, or psychological disorders that limit exercise or mobility
* Being in another supportive program
* Being in the very active category according to the "International Physical Activity Scale (IPAQ- Short Form)"
* Being a severity of more than 4 points according to the "Modified Borg Scale (MBS)"
* Being a score of 2 and above according to the "ECOG Performance Scale"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ- Short Form) | Baseline and 8th week
  It is used to evaluate physical activity. The form includes walking, moderate and vigorous activity, sitting categories. The total score includes the sum of time (minutes) and frequency (days).
National Cancer Institute (NCI) -CTCAE v5.0 Toxicity Criteria | Baseline and 8th week
  This scale was developed to evaluate the grading of chemotherapy-related peripheral neurotoxicity. It evaluates sensory and motor neuropathy between grades 1-5.
Cancer Fatigue Scale | Baseline and 8th week
  This scale was developed to evaluate the fatigue of cancer patients. It includes 15 questions and three sub-dimensions: Physical, Affective and Cognitive. The Likert type form is evaluated by giving points. Increasing scores received from the scale demonstrate a high level of fatigue.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy (EORTC QLQ-CIPN 20) | Baseline and 8th week
  This scale was developed to evaluate the effect of peripheral neuropathy on quality of life of cancer patients. It includes 20 questions and three sub-dimensions: Sensory, Motor and Autonomic. The Likert type form is evaluated by giving points. Increasing scores received from the scale demonstrate a high level of symptoms and problems related to peripheral neuropathy.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline and 8th week
  This Scale was developed to measure the quality of life of patients with cancer. It includes 30 questions and three sub-dimensions: Global health status, Functional, Symptom. High scores in the functional subscale indicate good/healthy functional status, high scores in the symptom subscale indicate high levels of symptoms and/or problems, and high scores in the global health status/quality of life subscale indicate good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Arikan, PhD, RN, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Konyaalti, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No